CLINICAL TRIAL: NCT00675103
Title: Multicenter, Open-Label, 24 Week Regimen of 8 mg Pegloticase i.v. in Symptomatic Gout Subjects Who Participated in Previous Studies of Pegloticase i.v.
Brief Title: Re-exposure Study of Pegloticase Intravenous (i.v.) in Symptomatic Gout Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Savient Pharmaceuticals (Industry)
Responsible Party: Chief Medical Officer, Savient Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0409
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Gout Refractory to Conventional Therapy
Keywords: Gout; Gouty Arthritis; Anti-Gout preparations
MeSH Terms: conditions — Gout; Arthritis, Gouty | interventions — Pegloticase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pegloticase (Experimental)
  Interventions: Drug: pegloticase 8 mg i.v.

INTERVENTIONS:
Drug: pegloticase 8 mg i.v. — pegloticase 8 mg i.v. every 2 weeks for 24 weeks

SUMMARY:
The purpose of the study is to evaluate the safety and clinical effect of re-exposure to a 24 week course of treatment of pegloticase i.v. in subjects whose last exposure to pegloticase i.v. was at least one year before study entry.

This study is limited to four study centers in the US.

ELIGIBILITY:
Inclusion Criteria:

* Previous treatment in studies of pegloticase i.v.
* Last exposure to pegloticase i.v. greater than one year prior to study entry
* Symptomatic gout
* Documented hyperuricemic (SUA ≥ 7 mg/dL)

Exclusion Criteria:

* Prior exposure to Elitek® (rasburicase)
* Unstable angina
* Uncontrolled arrhythmia or hypertension
* Non-compensated congestive heart failure
* End stage renal disease requiring dialysis
* Concomitant use of SUA lowering agents and use of other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Chicago- Dept. Biological Services, Chicago, Illinois
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Portland Rheumatology Clinic, L.L.C., Lake Oswego, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegloticase 8 mg Every 2 Wks
Started | 7
Completed | 4
Not Completed | 3
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pegloticase 8 mg Every 2 Wks
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Profile
Description: Number of participants reporting events
Time Frame: 6 months
Measure: Number; unit: Number of participants
Arm/Group | Pegloticase 8 mg Every 2 Wks
Number analyzed (Participants) | 7
Number of participants
  Adverse Events | 7
  Serious Adverse Events | 2

2. Secondary Outcome: Mean Plasma Uric Acid
Description: This endpoint assessed the change in mean PUA concentration from baseline after the first dose and after the third dose. Mean PUA was calculated from samples collected at 5 timepoints following each of those doses. For example, Mean PUA at Week 3 included 5 timepoints before dose 2 infusion.
Time Frame: Baseline, Week 3 and Week 7
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pegloticase 8 mg Every 2 Wks
Number analyzed (Participants) | 7
mg/dL
  Baseline | 8.5 (1.21)
  Week 3 | 4.0 (2.63)
  Week 7 | 7.7 (5.61)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pegloticase 8 mg Every 2 Wks
Serious Adverse Events (participants affected / at risk) | 2
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pegloticase 8 mg Every 2 Wks
Cellulitis (Infections and infestations) | 1/7 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1/7 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegloticase 8 mg Every 2 Wks (N=7)
Infusion-Related Reaction (General disorders) | 4 (7)
Fatigue (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Gout (flare) (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Nausea (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Diabete Mellitus Non-Insulin Dependent (Metabolism and nutrition disorders) | 1
Tremor (Nervous system disorders) | 1
New Tophus (Musculoskeletal and connective tissue disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Wound Drainage (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less